CLINICAL TRIAL: NCT04159545
Title: Journeys Towards Citizenship: How People Cured of Hepatitis C (HCV) Using Direct-Acting Antiviral (DAA) Drugs Progress in a New HCV-free World. Future Destinations
Brief Title: Future Destinations: Journeys Towards Citizenship
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, John Dillon, Professor, University of Dundee
Other Study IDs: 2-39-19
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Hepatitis C; Drug Use
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants treated with DAAs: Participants identified through the standard pathway of care as receiving Direct-Acting Antiviral (DAA) drugs to treat chronic hepatitis C with a history of problematic substance use.
  Participants will be interviewed on 3 occasions over the course of 2 years. Participants views, meanings and value of cure will be explored through semi-structured interviews.
  Participants will also complete quantitative questionnaires to measure changes in drug taking behaviours of drugs used and frequency (WHO ASSIST 3.0 Q2), Map social networks (SIM-AIRing), Measure wellbeing in terms of economic and social value (Short Warwick- Edinburgh Mental Wellbeing Scale (SWEMWBS) and financial inclusion, household income and employment data).
  Interventions: Other: Qualitative and quantitative interviews
- Control Group: Participants identified through the standard pathway of care as having HCV positive antibodies who spontaneously clear the infection.
  Participants will be interviewed on 3 occasions over the course of 2 years. Participants views, meanings and value of cure will be explored through semi-structured interviews.
  Participants will also complete quantitative questionnaires to measure changes in drug taking behaviours of drugs used and frequency (WHO ASSIST 3.0 Q2), Map social networks (SIM-AIRing), Measure wellbeing in terms of economic and social value (Short Warwick- Edinburgh Mental Wellbeing Scale (SWEMWBS) and financial inclusion, household income and employment data).
  Interventions: Other: Qualitative and quantitative interviews

INTERVENTIONS:
Other: Qualitative and quantitative interviews — Qualitative semi-structured interviews and quantitative questionnaires

SUMMARY:
Hepatitis C is a liver disease caused by the hepatitis C virus (HCV), if left untreated it can lead to chronic liver disease, cirrhosis and cancer. HCV is a blood borne virus, the key risk group for HCV infection are those who currently inject drugs, or have done in the past.

For many years the treatment of chronic HCV infection was based on therapies that had significant side effects, long treatment period and were between 50-70% effective, this impacted on patient acceptability and compliance. However, for those completing the treatment and undergoing this "personal trial" literature describes the transformative experience of HCV cure and how people took steps towards a "normal life" moving beyond substance use.

Recent advances in Direct-Acting Antiviral (DAA) medicines available to cure HCV have transformed treatment with shorter treatment periods, few side effects, ease of administration and improved efficacy. However, there is a potential paradox, in that the DAA-based regimes provide a reliable cure, for a large majority of patients, with a relatively small treatment burden, but may not be a "personal trial" and may have a lesser impact on rehabilitation and recovery from substance use.

The success of attempts of the group cured of HCV with DAAs, to progress down a recovery pathway and to resume activities thought of as being part of normal citizenship, are therefore unclear.

This study will examine the types of activities that people cured of HCV undertake and the success of their recovery pathway, post-treatment with DAAs over a two year follow-up period.

DETAILED DESCRIPTION:
This study uses an ethnographic case study approach using mixed methods to describe the journey towards citizenship of people cured of HCV with DAAs through their recovery from substance use. Qualitative and quantitative data will be collected from participants in a series of three interviews over the course of a two year period.

Qualitative data collated will describe the views and experiences of those in this specific social situation and examine how this narrative evolves.

Quantitative data (Substance use (WHO ASSIST 3.0 Q2), Social Identity mapping, Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS), Participant capture form data - financial inclusion, household income and employment data) will be collected to demonstrate a physical quantifiable change to allow for data triangulation to describe the phenomenon under study.

The ethnographic case study will be delivered through the immersion of a qualitative researcher within the context of a community centre providing care for people who use drugs.

Case Setting

The Cairn Centre in Dundee is a partnership with Hillcrest, NHS Tayside, Dundee City Council and other voluntary sector partners. The centre is placed at the heart of the community in Dundee City and acts as an interface between people who inject drugs and the agencies that are established to support them. The Cairn centre offers a drop-in recovery cafe run by volunteers, providing a warm and welcoming environment for anyone interested in recovery. The atmosphere allows informal support for people with their recovery and a chance to socialise and meet other people in recovery. The centre also provides a backdrop for a variety of other sources of support available including drug and alcohol treatment, Blood Borne Virus testing and treatment, dentistry, ophthalmology, sexual health service, Keep Well Health checks, welfare and legal advice, housing and homeless advice, families mutual aid, overdose prevention training and naloxone as well as a variety of recovery groups helping people develop new skills and interests.

The Cairn centre is Dundee's busiest injecting equipment provision (IEP) provider and provides support and advice to active drug users as well as those in more advanced stages of recovery.

This study will also utilise other locations to capture the views of others who may not visit this setting. Utilising other locations adds to the validity of the study to capture the universe of experiences of those with problematic substance use treated with direct-acting antivirals and recognises that as people progress along a recovery journey their social setting may change. Other locations include drop-in services, hubs and Recovery Cafes run by third sector partners within Dundee, Angus and Perth & Kinross Health and Social Care Partnerships. NHS Tayside locations that provide drug services and community pharmacy contractors will also be utilised as locations.

Ethnographic case study Development of semi-structured interviews. An inductive approach will be taken to develop semi-structured interviews. A cohort of participants will be interviewed using broad, open interviews to explore the universe of experiences of this participant group in relation to substance use, testing and/or treatment of hepatitis C with direct acting-antivirals and life circumstances.

Themes will be explored until there is a consensus and no new emerging themes are identified. Explicit and Implicit emergent themes from the inductive interviews will be explored and evaluated by the researcher with triangulation within the research team alongside the literature and evidence of the theoretical frameworks "Recovery Capital" and "Identity Theories" to generate qualitative research questions. The qualitative research questions will be further explored by developing semi-structured interviews around the themes identified.

Researcher observation field notes The researcher will record participant observations during the interviews to provide rich verbatim descriptions of the specific situations, events and behaviours of the participants.

Thematic Analysis Thematic analysis will be used to identify, analyse and report patterns (themes) within the data using the computer assisted qualitative data analysis package NVivo.

The coding strategy will be open and emergent to allow new and emerging themes to be captured accurately.

Researcher triangulation of themes and coding strategy will be used to validate themes and minimise researcher bias. Cohen's Kappa coefficient will be reported at each stage to assess interpreter agreement.

After each interview and observation stage themes identified by the research team will be validated with participants to check the interpretation captured both implicit and explicit meanings of the pervious interview. This will be carried out at the end of the interview to minimise recall bias and influence of current interview stage answers.

The narrative and connecting analysis completed after the second interview stage will allow for a theory to be generated describing an authentic and accurate narrative of the personal value of cure of Hepatitis C. This theory will be tested at the final interview stage to allow for causal validation using the approaches of modus operandi and searching for negative cases.

Quantitative data collection Participant Capture Form Participant data will be collected at baseline, 2nd visit and 3rd visit to record age, gender, ethnic background, financial inclusion, household income and employment data, current and/or previous treatment for problematic substance use and any previous history of hepatitis C infection. Baseline is defined in this study as first visit after consent is given. Questions that cannot change will only be asked at baseline, for example ethnic origin.

Participants will be asked questions to identify demographics to ensure participants are purposively selected to describe the universe of themes and experiences.

The questions included are part of the Scottish Survey Core Questions and are recommended for use in other surveys due to:

* Comparability across surveys is improved
* Thoroughly tested questions to provide confidence that participants understand what is being asked
* Questions have been widely consulted on to reduce risk of offence when asking questions about a sensitive subject The researcher will assist the participant to complete these questions. Participants may decline to answer these questions if they find the subject difficult or embarrassing, in this event this will be recorded.

World Health Organisation Alcohol, Smoking and Substance Involvement Screening Test (WHO ASSIST 3.0) The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) was developed for the World Health Organization (WHO) to detect and manage substance use and related problems in primary and general medical care settings. This study will utilise Question 2 of the WHO ASSIST screening tool to provide a measure of substances used and frequency within the last three months. The question uses a 5 point Likert scale to provide a quantitative measure of substance use at that point in time. The participant will complete this form with the assistance of the researcher if required.

Social Identity Map- Ascertaining identity resources (SIM - AIRing) The participants will be asked to place their social networks on a mapping tool that will provide a graphic representation of the social network at that point in time. The participants name will not be recorded on the map, only the participant ID number. The map will demonstrate the number of social contacts within the network, a measure of the relationship (inner circle, outer circle and influence) and the substance use status of the members of the network. Participants will be asked to assign pseudo identities for their social network members. The pseudo identity is known only to the participant and will be insufficient for the researcher to identify an actual person.

The participant will rate the importance of their social network members (indicated by placing them in the inner or outer circle) and indicate their status as user, non-user or in recovery. Social contact pseudo identities will be assigned coloured dots to indicate their status: red for active user, green for non-user and blue for individuals in recovery. This tool provides a quantitative measure of social network and will be mapped at each interview stage so that longitudinal insights into the change in social influences may be clearly described.

The researcher will assist the participant to complete this map.

Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) Participants will be asked to complete the self-reported short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) with assistance from the researcher if required. The measure is a list of 7 positive mental health statements with 5 response categories assigned scores and the total scores calculated. Movements in the total wellbeing score have been valuated using the wellbeing valuation method and represent the additional money the average individual would need to improve their wellbeing, which is the same as the improvement in their SWEMWBS score. This measurement can then be used to calculate a social value impact.

Data collection A baseline measure of patient demographics will be recorded at the first interview stage and at each interview to describe any changes over time.

Participants will be followed over a 2 year interval with an aim of 3 contacts over that period. Interviews at baseline and followed up between 6-18 months after baseline and at the end point over a 2 year period. Qualitative and Quantitative data will be collected and analysed at each interview stage.

A narrative of the final destinations achieved for those cured of HCV using DAAs will be reported with a description of how this cure changes participant's perspectives on their place in society, a personal value of a cure and changes in social network structures.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a history of problematic substance use with chronic HCV infection who are or have been treated with DAAs.
* Adults who have a history of problematic substance use and positive HCV antibodies who spontaneously clear the infection (control group)
* People of any ethnic origin who are able to speak English and are willing to talk about and reflect on their experiences with the phenomenon under study.
* Participants willing to have the semi-structured interviews audio recorded.

Exclusion Criteria:

* Participants with no history of problematic substance use.
* Participants who are not willing to consent to the study
* Participants who do not speak English.
* Females who report being pregnant at the beginning if the study will be excluded.
* Females who become pregnant during the study period will be excluded, however data obtained prior to the pregnancy may still be included.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People with a history of problematic substance use and chronic hepatitis C infection prior or after treatment with DAAs or a control group with positive HCV antibodies who spontaneously clear the virus identified during standard pathway of care.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Non-clinical future destinations achieved | 2 years
  The views, meaning and value of cure for individuals cured of HCV with DAA's and the non-clinical future destinations achieved.

SECONDARY OUTCOMES:
Measurement in drug taking behaviours of drugs used and frequency | 2 years
  WHO ASSIST 3.0 Q2 questionnaire
Map of social network with a measure of individuals with problematic substance use, those in recovery and those with no history of problematic substance use. Measuring changes over the time frame. | 2 years
  Social Identity mapping - Ascertaining Identity Resources (SIM-AIRing)
Measure, understand and communicate the economic and social value of the non-clinical outcomes of potential changes of those cured of HCV with DAAs | 2 years
  Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) and financial inclusion, household income and employment patient demographic capture form

CONTACTS AND LOCATIONS:
Overall Officials: Sarah R Donaldson, MPharmS, Principal Investigator — University of Dundee
Locations (1):
- Cairn Centre, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: No